CLINICAL TRIAL: NCT01388816
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate Efficacy, Safety and Tolerability of DRL-17822 in Patients With Type II Hyperlipidemia
Brief Title: A Safety and Efficacy Study of DRL-17822, a Cholesteryl Ester Transfer Protein (CETP) Inhibitor, in Patients With Abnormal Cholesterol Levels
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Collaborators: PharmaNet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRL-17822/CD/004
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Results first posted 2014-04-22 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-03

CONDITIONS: Type II Hyperlipidemia
Keywords: Randomized; Double-Blind; Placebo Controlled; Parallel Arm; Type II Hyperlipidemia; Cholesteryl Ester Transferase Protein Inhibitor; CETP Inhibitor
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — DRL-17822

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo capsule (Placebo Comparator)
  Interventions: Drug: DRL-17822 or placebo
- DRL-17822 50 mg (Experimental)
  Interventions: Drug: DRL-17822 or placebo
- DRL-17822 150 mg (Experimental)
  Interventions: Drug: DRL-17822 or placebo
- DRL-17822 300 mg (Experimental)
  Interventions: Drug: DRL-17822 or placebo

INTERVENTIONS:
Drug: DRL-17822 or placebo — DRL-17822 50, 150 or 300 mg or matching placebo once daily after breakfast

SUMMARY:
The purpose of this study is to determine if a new drug, DRL-17822, is safe and effective in elevating high density lipoprotein cholesterol (HDL-C) and reducing low density lipoprotein cholesterol (LDL-C) in people with abnormal cholesterol levels that may put them at risk for heart disease.

DETAILED DESCRIPTION:
Cardiovascular disease is a leading cause of death worldwide. Among cardiovascular disorders, coronary heart disease (CHD) caused by atherosclerosis is the most common cause of morbidity and mortality. Prevention, stabilization and regression of atherosclerotic plaques may have a major impact on reducing the risk of acute coronary events.

LDL-C lowering agents, primarily the statins, are the current mainstay in the pharmacologic management of dyslipidemia. However even with stain use, residual CHD risk from dyslipidemia remains. Epidemiologic and observational studies have shown that HDL-C is also a strong independent predictor of CHD, suggesting that raising HDL-C levels might afford clinical benefit in the reduction of cardiovascular risk.

Presently only niacin is approved by the FDA for HDL-C elevation and can raise HDL-C levels by 20-30%. However its use can be limited by a high incidence of flushing and, less commonly, by elevation of blood glucose and potential hepatic toxicity.

Cholesteryl ester transfer protein (CETP) inhibitors are being explored for their ability to elevate HDL-C. A small molecule CETP inhibitor, torcetrapib, has been demonstrated to elevate HDL-C by 60-100%. However, a large clinical trial (ILLUMINATE) where it increased HDL-C by a mean of 72% compared to baseline was halted as it failed to show benefit. Post-hoc analysis of this study implicated an off-target increase in blood pressure as potentially counteracting any anti-atherosclerotic benefits. Post-hoc subgroup analysis showed that patients in the highest HDL-C quartile had a 57% reduction in the risk of cardiovascular events.

Increased blood pressure appears to be specifically related to torcetrapib as two other small molecule CETP inhibitors, anacetrapib and dalcetrapib, have not shown this in clinical trials and have been well tolerated. DRL-17822 has also not shown elevation of blood pressure in either animals or in normal volunteers.

This study will investigate the efficacy and tolerability of DRL-17822 as dyslipidemia monotherapy in patients with Type II hyperlipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type II hyperlipidemia having lipid values of HDL-C: males ≤ 44 mg/dL (≤1.13 mmol/L), females ≤ 54 mg/dL (≤1.39 mmol/L); LDL-C: ≥ 130 mg/dL (≥3.33 mmol/L);
* Male or female, 18 to 70 years of age, inclusive. Female patients must be postmenopausal or surgically sterile. Men, unless surgically sterile must practice birth control from screening until the end of the study;
* Ability and willingness to give written informed consent;
* No clinically significant abnormal findings on medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory profiles of both blood and urine.

Exclusion Criteria:

* Patients with significant cardiac disease such as myocardial infarction, heart failure, coronary or peripheral artery angioplasty, bypass graft surgery, severe or unstable angina pectoris, cardiac arrhythmias, hypertension or any other disease which requires treatment;
* Uncontrolled diabetes (HbA1c > 8.0%);
* History of symptomatic cerebrovascular disease such as symptomatic carotid artery disease, cerebrovascular hemorrhage, transient ischemic attack or carotid endarterectomy or any disease which requires treatment;
* History of clinically significant hematologic, renal, hepatic, neurologic, endocrine, oncologic, pulmonary, immunologic or psychiatric disorders;
* Any current or recent (within 4 weeks of run-in) concomitant therapy (apart from paracetamol/acetaminophen and non-steroidal anti-inflammatory drugs [NSAIDs]). Patients on previous concomitant treatment may enter the study if the treatment has been discontinued, when appropriate and if ethically justified, at least four weeks prior to run-in;
* Body mass index (BMI)> 35 kg/m(2);
* Positive for hepatitis B, C or HIV or known history or concurrent tuberculosis;
* Positive drug screen result (i.e., cocaine, opiates, amphetamine, cannabis, barbiturates, benzodiazepines and/or metadone);
* Pregnant, breast feeding or women of child-bearing potential;
* Regular use of non-drug therapies such as garlic supplements and St. John's Wort;
* Presence or history of alcoholism or drug abuse;
* Use of more than 21 units of alcohol per week for males or more than 14 units per week for females;
* Smoking within 3 months prior to screening;
* Relevant drug hypersensitivity or allergy or any serious adverse event reaction to lipid regulating agents;
* Administration of study drug in another drug study within 90 days prior to enrollment or participation in another drug trial from screening to last follow-up of this study; Any surgical or medical condition which makes the patient unsuitable to participate in the opinion of the Investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2011-07; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kent Allenby, MD, Study Director — Dr. Reddy's Laboratories
Locations (12):
- Italy (5):
  - Genova
  - Milan
  - Modena
  - Palermo
  - Perugia
- Poland (4):
  - Gdynia
  - Gniewkowo
  - Katowice
  - Wroclaw
- Ukraine (3):
  - Chernivtsi
  - Kharkiv
  - Kyiv

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo; DRL-17822 50 mg; DRL-17822 150 mg; DRL-17822 300 mg: Once daily after breakfast
Period: Overall Study
Arm/Group | Placebo | DRL-17822 50 mg | DRL-17822 150 mg | DRL-17822 300 mg
Started | 45 | 43 | 44 | 44
Completed | 43 | 39 | 41 | 44
Not Completed | 2 | 4 | 3 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Placebo Capsule; DRL-17822 50 mg; DRL-17822 150 mg; DRL-17822 300 mg: Once daily after breakfast
- Total: Total of all reporting groups
Arm/Group | Placebo Capsule | DRL-17822 50 mg | DRL-17822 150 mg | DRL-17822 300 mg | Total
Number analyzed (Participants) | 45 | 43 | 44 | 44 | 176
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.0 (8.49) | 55.8 (9.93) | 54.2 (10.48) | 56.2 (10.74) | 55.8 (9.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 26 | 19 | 26 | 99
  Male | 17 | 17 | 25 | 18 | 77
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 45 | 43 | 43 | 44 | 175
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in HDL-C From Baseline
Description: Percent change from baseline in HDL-C after 28 days of treatment in patients with Type II hyperlipidemia
Time Frame: 28 days
Population: Intention to treat (ITT) analysis with last observation carried forward (LOCF) for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Placebo Capsule | DRL-17822 50 mg | DRL-17822 150 mg | DRL-17822 300 mg
Number analyzed (Participants) | 44 | 42 | 43 | 44
percent change from baseline | 3.2 (16.723) [-10.8 to 17.3] | 84.2 (42.000) [69.8 to 98.6] | 122.1 (60.035) [107.8 to 136.3] | 160.6 (57.325) [146.5 to 174.6]

2. Secondary Outcome: Safety and Tolerability of DRL-17822
Description: Incidence of treatment-related adverse events
Time Frame: 28 days
Population: Safety/ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo Capsule | DRL-17822 50 mg | DRL-17822 150 mg | DRL-17822 300 mg
Number analyzed (Participants) | 45 | 43 | 43 | 44
participants
  Treatment-related AEs | 4 | 3 | 3 | 4
  Severe AEs | 1 | 1 | 0 | 0

3. Secondary Outcome: Changes in Vital Signs Including Blood Pressure
Description: Vital sign abnormalities reported as treatment-emergent AEs
Time Frame: 28 days
Population: ITT/Safety Population
Measure: Number; unit: participants
Arm/Group | Placebo Capsule | DRL-17822 50 mg | DRL-17822 150 mg | DRL-17822 300 mg
Number analyzed (Participants) | 45 | 43 | 43 | 44
participants | 2 | 1 | 1 | 2

4. Secondary Outcome: To Evaluate Trough Levels of DRL-17822 in Plasma
Description: Trough levels of DRL-17822 in plasma after 28 days of treatment
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DRL-17822 50 mg | DRL-17822 150 mg | DRL-17822 300 mg
Number analyzed (Participants) | 40 | 41 | 44
ng/mL | 315.6 (227.2) | 826.2 (1124.6) | 1341.3 (1121.5)

5. Secondary Outcome: Changes in CETP Inhibition in Plasma
Description: Percent change from baseline in CETP Inhibition
Time Frame: 28 days
Population: ITT with LOCF
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage from baseline
Arm/Group | Placebo Capsule | DRL-17822 50 mg | DRL-17822 150 mg | DRL-17822 300 mg
Number analyzed (Participants) | 44 | 42 | 43 | 44
percentage from baseline | 7.2 [0.3 to 14.1] | 60.5 [53.4 to 67.6] | 79.7 [72.6 to 86.8] | 82.0 [75.2 to 88.9]

6. Secondary Outcome: Changes in Other Lipids and Apolipoproteins
Description: Change from baseline (LOCF, ITT population)
Time Frame: 28 days
Population: ITT with LOCF
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage change from baseline
Arm/Group | Placebo Capsule | DRL-17822 50 mg | DRL-17822 150 mg | DRL-17822 300 mg
Number analyzed (Participants) | 44 | 42 | 43 | 44
percentage change from baseline
  LDL-C | 4.9 [-5.8 to 15.5] | -15.4 [-26.3 to -4.5] | -18.7 [-29.5 to -7.9] | -39.4 [-50.1 to -28.8]
  HDL-C/LDL-C Ratio | 0.6 [-41.2 to 42.3] | 140.6 [97.9 to 183.3] | 240.0 [197.8 to 282.2] | 385.2 [343.5 to 427.0]
  Total Cholesterol | 1.5 [-2.9 to 5.8] | -0.9 [-5.3 to 3.5] | -0.8 [-5.2 to 3.5] | -0.8 [-5.1 to 3.5]
  Triglycerides | 4.5 [-7.7 to 16.7] | -14.2 [-26.7 to -1.7] | 0.9 [-11.5 to 13.2] | -11.3 [-23.5 to 1.0]
  Apo A1 | 1.8 [-4.1 to 7.7] | 35.0 [29.0 to 41.1] | 44.8 [38.8 to 50.8] | 59.1 [53.2 to 65.1]
  Apo B | 2.9 [-2.4 to 8.2] | -15.1 [-20.5 to -9.7] | -22.2 [-27.6 to -16.9] | -28.9 [-34.2 to -23.6]
  Apo E | 3.9 [-13.7 to 21.4] | 2.6 [-15.3 to 20.6] | 10.9 [-6.9 to 28.6] | 32.5 [15.0 to 50.1]
  Apo Lp(a) | 2.8 [-34.4 to 40.0] | -26.2 [-63.9 to 11.4] | 10.0 [-26.2 to 46.2] | -37.7 [-75.4 to -0.1]

ADVERSE EVENTS:
Time Frame: From randomization to 28 days of treatment
Arm/Group | Placebo Capsule | DRL-17822 50 mg | DRL-17822 150 mg | DRL-17822 300 mg
Serious Adverse Events (participants affected / at risk) | 1/45 | 1/43 | 0/43 | 0/44
Other Adverse Events (participants affected / at risk) | 8/45 | 4/43 | 6/43 | 2/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Capsule (N=45) | DRL-17822 50 mg (N=43) | DRL-17822 150 mg (N=43) | DRL-17822 300 mg (N=44)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Pericecal abscess treated with antibiotic therapy
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Treated as an outpatient
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Capsule (N=45) | DRL-17822 50 mg (N=43) | DRL-17822 150 mg (N=43) | DRL-17822 300 mg (N=44)
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 2
Pyrexia (Investigations) | 1 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 3 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less